CLINICAL TRIAL: NCT03349684
Title: A Multicenter, Randomized, Double-Blinded, Monotherapy-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of the Acarbose and Metformin in Loose-Dose Combination Compared to Metformin Monotherapy in Subjects WithType 2 Diabetic Mellitus (T2DM) That is Inadequately Controlled by Metformin Monotherapy
Brief Title: Loose-dose Combination of Acarbose and Metformin for T2DM in Metformin-failure Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17886
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acarbose plus metformin arm (Experimental): Participants received loose combination of acarbose and metformin 3 times daily.
  Interventions: Drug: Acarbose; Drug: Metformin; Drug: Placebo
- Metformin plus placebo arm (Active Comparator): Participants received loose combination of placebo and metformin 3 times daily.
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Acarbose — Uptitrated in the treatment phase from 50 mg per day for 1 week, followed by 100 mg per day for another week, and 150 mg per day for the rest 14 weeks, oral, with the first mouthful of main meal
  Arms: Acarbose plus metformin arm
Drug: Metformin — 500 mg 3 times daily, oral, with the first mouthful of main meal
Drug: Placebo — Acarbose matching placebo, oral

SUMMARY:
To demonstrate the efficacy and safety of acarbose and metformin loose-dose combination as compared to metformin monotherapy in the treatment of subjects with T2DM that is inadequately controlled by metformin alone

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 18 to less than 80 years
* Diabetes mellitus type 2, that is insufficently controlled with metformin defined by HbA1c between 7.0 % and 10.0%, inclusive
* Body mass index between 22 and 45 kg/m^2, inclusive
* Women and men of reproductive potential must agree to use adequate contraception when sexually active

Exclusion Criteria:

* Fasting plasma glucose > 14.0 mmol/L
* Severe metabolic diabetic complications

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Absolute change in the levels of glycosylated hemoglobin (HbA1c) | At baseline and at treatment week 16

SECONDARY OUTCOMES:
Responder rates | At week 16
  Defined as the percentage of subjects who achieve optimal glycemic control, defined by hemoglobin A1c of 1) < 7%, and 2) < 6.5%
Change in 2-hour postprandial plasma glucose (PPG) | At baseline and at treatment week 16
Change in fasting plasma glucose (FPG) levels | At baseline and at treatment week 16
Change in fasting serum insulin levels | At baseline and at treatment week 16
Change in insulin resistance score | At baseline and at treatment week 16
  Insulin resistance score was calculated based on the homeostasis model assessment (HOMA) model: fasting plasma glucose in mmol/l * fasting serum insulin in mU/L / 22.5.
Number of participants with adverse events | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (29):
- China (29):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hosp. Sun Yat-Sen Univ., Guangzhou, Guangdong
  - The 3rd Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affliated Hospital of Hainan Medical University, Haikou, Hainan
  - Hainan Third People's Hospital (Province Nongken Sanya Hopt), Sanya, Hainan
  - 1st Affiliated Hospital of Henan Science and Technology Univ, Luoyang, Henan
  - The first affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - Tongji Hosp. of Tongji Med Coll, Huazhong Uni of Sci & Tech., Wuhan, Hubei
  - Chenzhou No. 1 People's Hospital, Chenzhou, Hunan
  - 1st Peopl's Hosp of Changzhou 3rd Affil Hosp of Soochow Univ, Changzhou, Jiangsu
  - Huai'an First People's Hospital, Nanjing Medical University, Huai'an, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jilin Province People's Hospital, Changchun, Jilin
  - 1st Affiliated Hospital of Xi'an Jiaotong Medical University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Emergency General Hospital, Beijing
  - Peking Union Medical College Hospital CAMS, Beijing
  - Beijing Pinggu Hospital, Beijing
  - Changsha Central Hospital, Changsha
  - Jiangxi PingXiang people's Hospital, Pingxiang
  - Shanghai Tenth People's Hospital, Shanghai
  - Tianjin Union Medicine Centre (People's Hospital of Tianjin), Tianjin